CLINICAL TRIAL: NCT04818554
Title: Epidemiology and Prognosis of ARDS After Pulmonary Resection Surgery
Acronym: ARDS_THO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0191
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Thoracic; Pulmonary Restrictive Disease; ARDS
Keywords: Thoracic surgery; ARDS; Pulmonary resection; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The improvement in ARDS mortality over the last 20 years seems to be largely explained by the reduction of mechanical ventilation-induced injury (VILI). VILI is essentially related to volotrauma closely associated with "strain" and "stress". The pulmonary stress corresponds to the transpulmonary pressure (alveolar pressure - pleural pressure), and the strain to the change in lung volume related to the functional residual capacity (FRC) of the injured lung at PEEP = 0. The volotrauma corresponds therefore to the generalized excess of stress and strain on the injured lung.

The initial therapeutic strategy consists in protective ventilation with a tidal volume of 6 ml/kg of theoretical ideal weight (predicted by height), associated with a high respiratory rate between 25 and 30 cycles per minute to control PaCO2 (< 50 mmHg), apply a high positive expiratory pressure PEEP according to FiO2, maintain a plateau pressure (PP) lower than 30 cmH20, reduce instrumental dead space, use curarization, recruitment maneuvers such as alternate prone, improve ventilation-perfusion adequacy using inhaled NO.

As a last resort, extracorporeal oxygenation by veno-venous ECMO is a device to supplement respiratory function by improving oxygenation and ensuring decarboxylation. Veno-venous ECMO is indicated in severe ARDS with PaO2/FiO2 < 80 mmHg and/or when mechanical ventilation becomes unsafe due to increased plateau pressure despite optimized ARDS management including high PEEP levels, curarization and prone position.

After lung resection surgery, the incidence of ARDS is 2-8% and its prognosis remains more poor, despite advances in management, with a mortality of up to 60%. Risk factors include intraoperative vascular filling, type of pulmonary resection, and predicted postoperative respiratory function. Early support with VV ECMO is vital in some patients to treat severe hypoxemia, due to variable surgical reduction of lung parenchyma depending on carcinological involvement or initial lung pathology. ). There are very few data concerning these patients with pulmonary resection. The primary objective of this study is to describe the prevalence of ARDS and the risk factors for its occurrence after pulmonary resection surgery. The secondary objective is to compare the ventilation parameters (especially motor pressure) in patients with reduced lung parenchyma in ARDS under VV ECMO with those who did not use VV ECMO assistance.

ELIGIBILITY:
Inclusion criteria:

- Patient hospitalized following ARDS after thoracic resection surgery

Exclusion criteria:

- Refusal to participate after receiving the information letter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ARDS hospitalized in the DAR ADV intensive care unit after thoracic resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ARDS | 1 day
  Prevalence of ARDS after pulmonary resection surgery
risk factors for its occurrence after pulmonary resection surgery | 1 day
  risk factors for its occurrence after pulmonary resection surgery

SECONDARY OUTCOMES:
According to the usual clinico-biological data of monitoring in intensive care | 1 day
  According to the usual clinico-biological data of monitoring in intensive care

CONTACTS AND LOCATIONS:
Overall Officials: hélène David, PHD, Study Director — UH MONTPELLIER
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC